CLINICAL TRIAL: NCT03504098
Title: Folate One-carbon Malnutrition as the Metabostemness Risk Factor of Malignancy Tumor Development and the Prognostic Predictor of Non-small Cell Lung Cancer Patients
Brief Title: Folate One-carbon Malnutrition as the Metabostemness Risk Factor of Malignancy Tumor Development of NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201701123RINC
Record Dates: First submitted 2018-03-25; First posted 2018-04-20 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: One-carbon metabolism; Folate; Choline; metabolomic marker; Cancer risk
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample 10c.c
  lung tumor tissue
  non-lung tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lung cancer patients tumor: Using to analysis metabolomic markers, one carbon folate nutrition levels in lung cancer patients.
- Lung cancer patients blood: Using to analysis folate, B12, homocysteine levels in plasma and RBC. Using to analysis cDNA gene test in buffy coat.
  Interventions: Behavioral: nutrition consult
- Lung cancer patients: Supply nutrition counseling
  Interventions: Behavioral: nutrition consult

INTERVENTIONS:
Behavioral: nutrition consult — Post-lung cancer operation diet pattern
  Groups: Lung cancer patients; Lung cancer patients blood

SUMMARY:
Non-small cell lung cancer (NSCLC) accounts for more than two-thirds of lung cancer, which is the leading cause of cancer deaths in Taiwan. The overall prognosis of NSCLC is poor with low 5-year survival rates. Recent advances suggest that malignancy NSCLC cancers are the cancer stem cell (CSC) diseases. The stemness potentials of CSC with epithelial-mesenchymal transdifferentiation ensure their invasion and disseminate to metastsis organs. The self-renewal property of CSC mediates intrinsic drug resistance to cytotoxicity therapy and promoted aggressive relapse tumour. Metabolic reprogramming on bioenergetics of malignant cancer cells has been proposed as the key mediator in the stemness CSC development. Malignancy cells uptake glucose for fermented glycolysis to produce lactate which release resulted in acidified microenvironment to trigger the mTOR and sonic hedgehog metabolic stress signaling in supporting CSC stemness potentials. The metabostemness of cancer cells is the new-dimensional hallmark of malignancy tumour, which may serve as the diagnostic markers for the early detection of malignancy cancers. Folate-mediated one carbon metabolism coordinates glucose into amino acid metabolism to tailor the fuel metabolites in supporting macromolecule synthesis and to sustain the bioenergetics requirement. Acting as the metabolic stressor, low folate intake is associated with increased risks of lung cancers. Folate and one-carbon nutrient status of NSCLC patients in Taiwan, however, has not been assessed. The role of low folate metabolic stress (LFMS) in metabostemness marker and metastasis potentials of malignancy NSCLC is unexplored. The causal effect and the working mechanisms by which LFMS promoted NSCLC malignancy remain elusive.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon diagnosed as the first time having non-small cell lung cancer from the surgical clinic of National Taiwan University Hospital

Exclusion Criteria:

* Patients Suffer from major diseases such as heart, liver, kidney, or peripheral arterial disease, or having mental illness
* Diabetes and non-lung cancer patients
* Pregnancy, breast-feeding pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who was diagnosed as the first time having NSCLC from NTUH. Patients have no chronic disease / other cancer / chemotherapy / radiotherapy. Patients at least 20 years old.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of one-carbon nutrient (folate, choline, betaine, Vitamine B12) intake of lung cancer patients | Past 0.5-1 year
  Using semiquantitative food frequency questionnaires

SECONDARY OUTCOMES:
Measure maternal blood biochemistry (folate, choline, betaine, homocysteine, Vitamine B2, Vitamine B6, Vitamine B12, etc.) | At baseline
  Using blood analysis to calculate the levels of one carbon nutrition
Assessment of one-carbon nutrient metabolomic markers in lung cancer patient tumor tissue | 3 years
  Using LC/MS or GC/MS to claculate metabolomic markers

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Pao Cheng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan